CLINICAL TRIAL: NCT03949426
Title: A First-in-Human, Randomized, Double-blind, Placebo-controlled, Sequential Parallel Group, Single Ascending Dose Study in Healthy Participants to Evaluate the Safety, Tolerability and Pharmacokinetics of KPG-818
Brief Title: Safety, Tolerability and Pharmacokinetics of KPG-818 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kangpu Biopharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KPG-818-SLE-101
Record Dates: First submitted 2019-05-08; First posted 2019-05-14 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: Parallel and Sequential
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study is double-blind with regard to treatment (KPG-818 or placebo) at each dose level. Any clinical staff involved in the preparation or administration of the study intervention and who are unblinded will take no further part in the study. will remain blinded during the study conduct, unless otherwise required based on study findings. The pharmacokineticist will be unblinded to perform the final PK analyses after all participants have completed the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KPG-818 (Experimental): Dose escalation
  Interventions: Drug: KPG-818
- Placebo (No Intervention): Matching placebo

INTERVENTIONS:
Drug: KPG-818 — KPG-818 Capsules (1 mg, 5 mg and 20 mg) for oral administration is the drug substance powder filled in capsule (PIC) dosage form. KPG-818 Capsules and placebo capsules are packaged in HDPE bottle capped with HDPE cap.
  Other Names: Matching placebo
  Arms: KPG-818

SUMMARY:
This is a Phase 1 study to investigate the safety, tolerability and pharmacokinetics (PK) of KPG-818 in healthy male and female participants and the effect of food on the PK of KPG-818. The study will assist in identifying appropriate, well tolerated doses that can be administered in subsequent studies in healthy participants and participants with systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
A total of 40 subjects will be evaluated with 30 subjects randomized to receive active drug and 10 subjects randomized to receive placebo in a double-blind fashion (8 subjects in each dose cohort, 6 subjects randomized to active drug and 2 subjects randomized to placebo). Five dose levels (2, 5, 10, 20 and 30 mg) are planned to be evaluated.The study will be double blinded with regard to treatment (KPG-818 or placebo) at each dose level. KPG-818 and placebo will be matched for formulation, appearance and number of capsules. Safety assessments will be performed throughout the study including physical examinations, vital signs, clinical laboratory tests, 12 lead electrocardiograms and monitoring of adverse events. Pharmacokinetic blood and urine samples will be collected up to 72 hours after dosing. A post-treatment follow-up visit will be performed within 10 days of the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all the following criteria apply:

1. Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
2. Participants who are healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and ECGs.
3. Body mass index (BMI) within the range 19 to 30 kg/m2 (inclusive).
4. Males and females of non-childbearing potential.
5. A male participant must agree to use a highly effective contraception as detailed in Appendix 4 of this protocol during the intervention period and for at least 3 months after the dose(s) of study intervention and refrain from freezing or donating sperm during this period and for 3 months after dosing.
6. A female participant is eligible to participate if she is not a woman of childbearing potential (WOCBP) as defined in Appendix 4. Female participants must have been surgically sterilized (bilateral oophorectomy or bilateral salpingectomy at least 3 months before the start of the study and/or hysterectomy); have premature ovarian failure confirmed by a specialist gynecologist; be postmenopausal (defined as ≥ 50 years and naturally [spontaneously] amenorrheic (postmenopausal) for ≥ 12 months); or have XY genotype, Turner syndrome or uterine agenesis.
7. Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

1. Participant has clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological or psychiatric disorder(s) as determined by the Investigator.
2. History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
3. Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of study intervention.
4. Any clinically important abnormalities in clinical chemistry, hematology or urinalysis results as judged by the Investigator, and confirmed by a repeat measurement at the Screening Visit or at admission (Day -1).
5. Any positive result at the Screening Visit for serum hepatitis B surface antigen, hepatitis C antibody and human immunodeficiency virus (HIV).
6. Abnormal vital signs, after 5 minutes supine rest, as judged by the Investigator to be clinically significant, and confirmed by a repeat measurement at the Screening Visit or at admission (Day -1).
7. Any history or presence of an abnormal ECG, which, in the Investigator's opinion, is clinically significant, confirmed by a repeat measurement at the Screening Visit or at admission (Day-1).
8. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to KPG-818.
9. Judgment by the Investigator that the participants should not participate in the study if they have any ongoing or recent (i.e., during the Screening Period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
10. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to administration of study intervention.
11. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to administration(s) of study intervention or longer if the medication has a long half-life.
12. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days or 5 half-lives, whichever is longer, of the first administration of study intervention in this study.
13. Known or suspected history of drug abuse as judged by the Investigator.
14. Current smokers or past smokers who have smoked or used nicotine products (including e-cigarettes) within the previous 3 months prior to the Screening Visit.
15. History of alcohol abuse or excessive intake of alcohol as judged by the Investigator.
16. Positive screen for drugs of abuse, alcohol or cotinine (nicotine) at the Screening Visit or admission to the Clinical Unit.
17. Participants who consume greater than 500 mg of caffeine or xanthine-containing products per day (e.g., coffee, tea, soft drinks, energy drinks, chocolate,) or who refuse to abstain from caffeine-containing or xanthine-containing foods or beverages from 48 hours prior to admission (Day -1) until discharge from the clinical unit.
18. Use of red wine, Seville oranges, grapefruit or grapefruit juice, pomelos, exotic citrus fruits, or grapefruit hybrids from 7 days before the start of study intervention (Day 1) in each dosing session (as applicable) until collection of the final PK sample in each dosing session (as applicable).
19. Use of alcohol within 72 hours of dosing (Day 1).
20. Participants who are vegans or have medical dietary restrictions.
21. Participants who cannot communicate reliably with the Investigator.
22. Vulnerable participants, e.g., kept in detention, protected adults under guardianship, trusteeship or committed to an institution by governmental or juridical order.
23. Involvement of any Kangpu Biopharmaceuticals, Ltd. or study site employee or their close relatives.
24. Plasma donation within 1 month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to the Screening Visit and for at least 3 months after the dose(s) of study intervention.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 72 hrs post-dose
  Number of Treatment-Emergent Adverse Events(TEAE)
Maximum Tolerated Dose [Safety and Tolerability] | Up to 72 hrs post-dose
  If dose escalation is stopped based on available safety data, the current dose level will be considered as the Minimum intolerable dose (MID). The dose just below the MID will be regarded as the MTD. If the dose escalation is stopped due to reaching exposure limit without dose limiting safety findings, the MTD cannot be determined.

SECONDARY OUTCOMES:
Blood KPG-818 concentrations | Up to 72 hrs post-dose
  Blood samples for analysis of KPG-818 and KPG-818H will be collected at pre-dose (within 30 minutes) and 0.5, 1, 2, 4, 6, 10, 12 and 18 hours post-dose on day 1; 24 and 36 hours post-dose on day 2; 48 hours post-dose on day 3 and 72 hours post-dose on day 4.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Yoon, MD, Principal Investigator — California Clinical Trials
Locations (1):
- California Clinical Trials Medical Group, Glendale, California, United States